CLINICAL TRIAL: NCT04754750
Title: Differences in Lipid and Cognitive Change Between One-month and 3-month Paliperidone Palmitate Treatment in Stable Schizophrenia
Brief Title: Differences in Schizophrenia With One-month and 3-month Paliperidone Palmitate Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Calo Psychiatric Center (Other)
Responsible Party: Principal Investigator, For-Wey Lung, Professor, Calo Psychiatric Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 100-046
Record Dates: First submitted 2021-01-27; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenics
Keywords: paliperidone palmitate; social function; cognitive function; quality of life
MeSH Terms: conditions — Social Adjustment | interventions — Paliperidone Palmitate

STUDY DESIGN:
Intervention Model Description: Total of 72 participants, including 41 men and 31 female, were received the PP1M three months. The stable participants were shifted to PP3M for one year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INVEGA Sustenna (Active Comparator): INVEGA Sustenna is a one month long-acting injection (PP1M)
  Interventions: Drug: Paliperidone Palmitate 156 MG/ML Prefilled Syringe [Invega]
- INVEGA Trinza (Active Comparator): INVEGA Trinza is a three month long-acting injection (PP3M)
  Interventions: Drug: Paliperidone Palmitate 546 MG Intramuscular Suspension, Extended Release [INVEGA TRINZA]

INTERVENTIONS:
Drug: Paliperidone Palmitate 156 MG/ML Prefilled Syringe [Invega]
  Other Names: Sustenna
  Arms: INVEGA Sustenna
Drug: Paliperidone Palmitate 546 MG Intramuscular Suspension, Extended Release [INVEGA TRINZA]
  Other Names: Trinza
  Arms: INVEGA Trinza

SUMMARY:
Schizophrenia is a chronic and severe psychiatric disorder, these patients suffer from positive symptoms, negative symptoms and cognitive deficits, of which working memory problems are considered a central cognitive impairment. Atypical antipsychotics are believed to have a superior effect in reducing both positive and negative symptoms of schizophrenia, coupled with a low risk of extrapyramidal symptoms. Particularly, 2nd-generation antipsychotic medications are commonly used in treatment of schizophrenia. An antipsychotic drug, Paliperidone palmitate (PDP), is administered to patients with schizophrenia as injections at one-month (PP1M) or three-month (PP3M) intervals. This study was compare the effects of treatment, social function, and side effects between PP1M and PP3M in patients with schizophrenia. Moreover, the changes of cognitive and lipid profile between two PDP were also explored. Firstly, participants were received the one month long-acting injection (PP1M) three months. Then, the stable participants were shifted to the three month long-acting injection (PP3M). Concomitant medications were allowed to prescribe except other antipsychotics. Outcome measurements were 20-item Toronto Alexithymia Scale (TAS-20), 45-itme quality of life for mental disorder (QOLMD), Short-version of the Udvalg for Kliniske Undersogelser (short-version UKU), and Wisconsin Card Sorting test (WCST). These measurements were performed every three-month except WCST which was performed every six-month. The different effects of PP1M and PP3M will be expected to find out in this study.

DETAILED DESCRIPTION:
This is a two and half-one years, single-arm, nonrandomized, open-label study which was conducted between Jan 2015 to Jun 2017 including from a psychiatric center in southern Taiwan. The stable schizophrenic patients who previously received risperidone long-acting injection for more than one year and shifted to paliperidone palmitate after including in the study. Firstly, participants were received the one month long-acting injection (PP1M) three months. Then, the stable participants were shifted to the three month long-acting injection (PP3M). Concomitant medications were allowed to prescribe except other antipsychotics. Outcome measurements were 20-item Toronto Alexithymia Scale (TAS-20), 45-itme quality of life for mental disorder (QOLMD), Short-version of the Udvalg for Kliniske Undersogelser (short-version UKU), and Wisconsin Card Sorting test (WCST). These measurements were performed every three-month except WCST which was performed every six-month. The effect of treatment was assessed using Personal and Social Performance (PSP) scales for the evaluation of psychosocial functioning at 0, 4, 8, and 12 weeks in first study, and at 0, 3, 6, 9, 12 months in second study, respectively. In addition, all participants were assessed for body weight, waist circumference, and blood lipid profile. To evaluate the lipid profiles, fasting blood samples were analyzed for total cholesterol (TC), Triglyceride (TG), High-density Lipoprotein (HDL) and Low-density Lipoprotein (LDL). These blood samples were collected at every month until study completion.

ELIGIBILITY:
Inclusion Criteria:

* All of them had to meet the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).

Exclusion Criteria:

* Patients who had comorbid serious medical illnesses, and may therefore present substantial clinical risk due to pharmacotherapy, were excluded from the sample, as were pregnant and lactating women.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Personal and Social Performance scales (PSP) | 15 months
  Personal and Social Performance scales was assessed for the evaluation of psychosocial functioning. A higher score represents better psychosocial functioning.
Short-version of the Udvalg for Kliniske Undersogelser (short-version UKU) | 15 months
  The Short-version of the Udvalg for Kliniske Undersogelser was assessed for the evaluation of psychic side effect. A higher score present to a mild or severe degree symptoms.
Wisconsin Card Sorting test (WCST) | 15 months
  Wisconsin Card Sorting Test was assessed for the performance of cognitive function. A higher score in conceptual level response and lower score in percent of perseverative errors present to greater cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: For-Wey Lung, MD, ScD, Principal Investigator — Calo Psychiatric Center

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04754750/Prot_SAP_000.pdf